CLINICAL TRIAL: NCT00907673
Title: The Automated Fluid Shunt (AFS)in Chronic Congestive Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovaShunt AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-CHF-001
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-12

CONDITIONS: Congestive Heart Failure; Ascites
MeSH Terms: conditions — Heart Failure; Ascites

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient condition pre-implant (Active Comparator)
  Interventions: Device: Automatic Fluid Shunt System

INTERVENTIONS:
Device: Automatic Fluid Shunt System — Fully implantable peritoneal catheter, bladder catheter, and pump
  Other Names: AFS System

SUMMARY:
A 28-week, feasibility study to investigate the safety and efficiency of the Automatic Fluid Shunt in patients with chronic congestive heart failure, ascites and diuretic resistance.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients ≥ 18 years of age
* A clinical diagnosis of chronic congestive heart failure > 6 months
* At least one episode of documented ADHF during the previous 6 months
* NYHA functional class III-IV
* Circulating levels of NT-proBNP ≥ 800 ng/L.
* Stable, optimized therapy for heart failure for at least 4 weeks prior to enrollment
* Echocardiography performed within 3 months
* Detectable ascites by ultrasound and/or computed tomography
* Diuretic resistance defined as a daily dose of furosemide > 80 mg, torsemide > 40 mg or bumetanide > 2 mg
* Written informed consent

Exclusion Criteria:

* Present or recurring systemic or local infection, such as peritonitis, urinary tract infection, or abdominal skin infection.
* Ongoing malignant disease with adverse prognosis
* Evidence of firmly loculated peritoneal effusion.
* Obstructive uropathy
* Severely reduced renal function (S-Creatinine 300 mol/l) or end-stage renal disease requiring dialysis
* Severe liver disease (ASAT and/or ALAT and/or total bilirubin three times upper limit of normal range laboratory values)
* Pregnancy
* Requirement for intravenous inotropes
* Acute coronary syndrome or any condition requiring emergency treatment
* Heart disease requiring surgical intervention during the course of the study
* Any other clinically significant disease that could be adversely affected by study participation judged by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To evaluate safety of the Automated Fluid Shunt device during a 28-week follow-up and to evaluate its efficacy by measuring change in NT-proBNP from baseline to 16 weeks, in patients with chronic congestive heart failure, ascites and diuretic resistance. | 16 and 28 weeks

SECONDARY OUTCOMES:
To determine the effect of AFS-treatment on functional capacity (NYHA class and 6-min. walking distance) compared from baseline to 16 and 28 weeks | 16 and 28 weeks
To determine change in LV volumes and LVEF (echocardiography) compared from baseline to 16 and 28 weeks | 16 and 28 weeks
To determine change in ascites, hydrothorax and leg edema (based on CT evaluation) compared from baseline to 16 and 28 weeks | 16 and 28 weeks
To determine change in renal function (GFR) compared from baseline to 16 and 28 weeks | 16 and 28 weeks
To determine change in quality of life based on Minnesota Living with Heart Failure Questionnaire (MLHFQ) compared from baseline to 4, 12 and 28 weeks | baseline to 4, 12 and 28 week

CONTACTS AND LOCATIONS:
Overall Officials: Kristjan Karason, MD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden